CLINICAL TRIAL: NCT00744198
Title: A Comparison in Terms of Efficacy and Safety Among Three Different Materials for Trans-obturator Correction of Urinary Stress Incontinence: Autologous, Synthetic and Biological Sling
Brief Title: Autologous Versus Synthetic Versus Biological Sling for Trans-obturator Correction of Urinary Stress Incontinence
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02/2008
Record Dates: First submitted 2008-08-26; First posted 2008-08-29 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Autologous; Biological; Mesh; Polypropylene; Sling; Synthetic; Stress incontinence; Surgery; TOT; Treatment
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (3):
- 1 (Active Comparator): Autologous sling
  Interventions: Procedure: Autologous transobturator tape procedure
- 2 (Active Comparator): Synthetic sling
  Interventions: Procedure: Synthetic transobturator tape procedure
- 3 (Active Comparator): Biological sling
  Interventions: Procedure: Biological transobturator tape procedure

INTERVENTIONS:
Procedure: Autologous transobturator tape procedure — A strip of rectus fascia is harvested. Small incision sites in the vagina and in the femoral/pelvic fold. Bilateral transobturator insertion of the autologous strip by means of reusable needles
  Arms: 1
Procedure: Synthetic transobturator tape procedure — Small incision sites in the vagina and in the femoral/pelvic fold. Bilateral transobturator insertion of synthetic mesh by means of mono-use needles.
  Arms: 2
Procedure: Biological transobturator tape procedure — Small incision sites in the vagina and in the femoral/pelvic fold. Bilateral transobturator insertion of biological mesh by means of mono-use needle
  Arms: 3

SUMMARY:
The treatment of urinary stress incontinence with trans-obturator approach, know as transobturatory tape (TOT), is a largely used sling-adopting procedures. The efficacy and safety of this minimally invasive surgery have been demonstrated, also in comparison with similar procedures, i.e transvaginal tape (TVT).

To date the results of TOT in terms of efficacy and safety described in literature mainly refer to procedure in which synthetic materials are used, whereas few data regarding the use of biological materials are available. Moreover, despite the well known benefits of the available synthetic and eterologue kit, their use may be limited by the high cost of these materials. At this proposal it can be suggested as alternative option the possibility to perform the procedure using an autologous tissue, i.e. rectus fascia, and reusable introductory needles. Based on these considerations the aim of this trial will be to compare autologous, synthetic and biological mesh for TOT in women with urinary stress incontinence.

DETAILED DESCRIPTION:
Women with genuine stress urinary incontinence will be enrolled and randomized in three groups (arm 1, arm 2, arm 3). All patients will be treated with a transobturatory approach, in patients of arm 1 will be used an autologous tissue and reusable introductory needles, in patients of arm 2 will be used a synthetic kit whereas in arm 3 will be a biological kit .

All eligible patients will undergo baseline assessment consisting of anthropometric, clinical, hormonal, urodynamic, and ultrasonographic evaluations. During the study, the surgical outcomes, the clinical subjective and objective efficacy data, and the adverse experiences will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Genuine stress urinary incontinence by self report, examination and test
* Urethral hypermobility
* Eligible for all three surgical procedures
* Ambulatory

Exclusion Criteria:

* Pregnancy
* <12 months post-partum
* Systemic disease and/or drugs known to affect bladder function
* Current chemotherapy or radiation therapy
* Urethral diverticulum, augmentation cytoplasty, or artificial sphincter
* Recent pelvic surgery
* Severe genuine stress incontinence (loss of urine with minimal physical activity) with associated prolapse equal to or more than second degree
* Previous pelvic or anti-incontinence surgery
* History of severe abdominopelvic infections
* Known extensive abdominopelvic adhesions
* Detrusor instability and/or intrinsic sphincter dysfunction
* Other gynaecologic pathologies (eg, fibroids, ovarian cysts)
* BMI >30

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 12 months

SECONDARY OUTCOMES:
Intra-operative complication rate | one day
Postoperative complications rate | 12 months
Failure rate | 12 months
Recurrence rate | 12 months
Quality of life | 12 months
Sexual function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Fulvio Zullo, MD, Study Chair — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Catanzaro, Italy